CLINICAL TRIAL: NCT05296668
Title: Cuffed Versus Uncuffed Tracheal Tubes in Neonates Undergoing Elective Surgery: a Double Blinded Randomized Controlled Trial
Brief Title: Cuffed Versus Uncuffed Tracheal Tubes in Neonates Undergoing Elective Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, Lecturer of Anesthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD-62-2021
Record Dates: First submitted 2022-03-17; First posted 2022-03-25 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Anesthesia, Endotracheal; Neonate
Keywords: Cuffed endotracheal tube; Neonates; General anesthesia

STUDY DESIGN:
Intervention Model Description: Recruited neonates will be randomly assigned to one of two groups in a 1:1 ratio; (group C) to receive a cuffed ETT and (group U) to receive an uncuffed ETT for airway management.
Who Masked: Participant, Outcomes Assessor
Masking Description: Induction of anesthesia will be performed by the attending senior anesthesia resident who has finished at least 2 years of residency (who is independent of the study team).
  All intraoperative measurements will be collected by an anesthetist who was not involved in the induction of anesthesia.
  All postoperative measurements will be collected by PACU nurse who is independent of the study team
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cuffed ETT group (Experimental): (group C) to receive a cuffed ETT for airway management.
  Interventions: Device: Cuffed ETT (Microcuff®, Halyard Health Inc., Atlanta, GA, USA); Device: Uncuffed ETT group
- Uncuffed ETT group (Active Comparator): (group U) to receive an uncuffed ETT for airway management.
  Interventions: Device: Cuffed ETT (Microcuff®, Halyard Health Inc., Atlanta, GA, USA); Device: Uncuffed ETT group

INTERVENTIONS:
Device: Cuffed ETT (Microcuff®, Halyard Health Inc., Atlanta, GA, USA) — (group C) to receive a cuffed ETT for airway management.
Device: Uncuffed ETT group — (group U) to receive an uncuffed ETT for airway management.
  Other Names: Uncuffed ETT (Mallinckrodt® Contour Murphy Eye)

SUMMARY:
This thesis aims to assess the safety and efficacy of usage of cuffed ETT in neonate undergoing elective surgeries.

DETAILED DESCRIPTION:
Neonates will be recruited into the trial during pre-operative assessment. Recruited neonates will be randomly assigned to one of two groups in a 1:1 ratio; (group C) to receive a cuffed ETT and (group U) to receive an uncuffed ETT for airway management. Randomization will be achieved using a computer-generated sequence. Concealment will be achieved using opaque envelopes.

All neonates will be anesthetized in accordance with the local policy of pediatric anesthesia unit in Abu El-Reesh pediatric hospital-Cairo university after ethics committee approval.

After preoperative examination and upon arrival to the operating room heart rate, noninvasive blood pressure NBP and oxygen saturation SPO2 will be monitored using standard monitor (drȁger infinity vista XL) before inhalational induction of anesthesia using titration of sevoflurane in oxygen air mixture 60% (starting from 3% up to 8%) until the neonate is put to sleep. Baseline lung ultrasound will then be done. After securing an intravenous line anesthesia will be completed with 1-2µg/kg of fentanyl and atracurium 0.5 mg/kg.

Induction of anesthesia will be performed by the attending senior anesthesia resident who has finished at least 2 years of residency (who is independent of the study team).

(Microcuff®, Halyard Health Inc., Atlanta, GA, USA), will be chosen for cuffed TTs, and (Mallinckrodt® Contour Murphy Eye) for non-cuffed tubes.

The appropriate ETT size will be decided by the attending anesthesia resident and will be based on the absence of resistance to insertion of the tube and the presence of audible leak (with inflation pressures of 20 cmH2O following initial cuff deflation for the cuffed ETT group). As necessary, ETT sizes will be adjusted one size up or down to achieve these conditions starting from 3mm internal diameter size.

For both groups: intubation trials will not exceed 2 times, or it will be excluded from the study.

Following inflation of the ETT cuff in C group, pressure will be measured using cuff manometry (Portex Limited, Hythe, Kent, UK) with cuff pressures will be monitored continuously, and if necessary, adjusted to pressures ≤ 20 cmH2O to allow for a good cuff seal without hyperinflation of the cuff.

Measurements will be carried out under both volume- controlled ventilation (VCV) and pressure-controlled ventilation (PCV) using (G.E-Datex-Ohmeda, Avance CS2, USA). Ventilation will be set initially to VCV of 6 ml/kg and PEEP 3 cmH2O. three anesthesia workstation measurements of inspiratory and expiratory tidal volumes will be recorded, and the mean taken for analysis of leakage around the ETT. Ventilation will then be adjusted to PCV of 10 cmH2O, PEEP of 3 cmH2O and leakage around the tube analyzed again in the same way. Then these measurements will be done again at 10 min and 20 min. Once these measurements are taken, ventilation will be continued as VCV of 6-8 ml/kg, PEEP 3 cmH2O and respiratory rate will be set between 30-40 to maintain end tidal CO2 within 30-40 mmHg for the remainder of the case.

At the end of the procedure and before return of spontaneous ventilation another set of measurements will be recorded.

In both groups, after return of spontaneous ventilation the neonates will be put on pressure support PS mode (PS 10, PEEP 3 and flow trigger of 1 L/min) and when the neonate is capable of triggering at least 70% of his own breathes and has good motor power; the ETT will be removed by the attending anesthetist after reversal of muscle relaxant effect using neostigmine 0.05 mg/kg with atropine 0.02 mg/kg and timing of extubation will be recorded.

All patients will be transported to the post anesthesia care unit PACU after ensuring that their airway and oxygenation are adequate. Oxygen saturation will be measured continuously until discharge from the PACU. Oxygen saturation will be recorded when the neonates are calm and the pulse oximeter showing consistent detection. Lowest measured SpO2 values will be recorded 10 min before removal of the ETT, and at 1 min, 5 min, 10 min, 15 min, 20 min and 30 min after removal.

Any respiratory adverse events (laryngospasm; bronchospasm; desaturation < 95%; airway obstruction; severe coughing and/or postoperative stridor) as well as subsequent interventions will be recorded and managed according to the local policy of Abo El Reesh pediatric hospital. All postoperative measurements will be collected by PACU nurse who is independent of the study team.

ELIGIBILITY:
Inclusion Criteria:

* • Neonates (infant in the first 28 days after birth)

  * Full term (more than 37 gestational weeks)
  * More than 3 kg bodyweight
  * ASA I-II
  * Scheduled for elective surgeries under general anesthesia requiring endotracheal intubation.

Exclusion Criteria:

* • Parents or legally authorized personnel refusal.

  * Anatomical abnormalities of upper air way.
  * Emergency surgery.
  * Low birth weight less than 3 kg
  * Surgery longer than 2 hours
  * Premature neonates
  * Upper airway surgery
  * Requirement for postoperative ventilation

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
The incidence of ETT exchange to find the appropriate ETT | 2 hours
  the incidence of ETT exchange to find the appropriate ETT defined as:(the absence of resistance to insertion of the tube and the presence of audible leak with inflation pressures of 20 cmH2O).

SECONDARY OUTCOMES:
Duration of intubation | 10 minutes
  calculated from time from the introduction of the laryngoscope blade to the mouth till the first trace of capnography recorded.
Leakage around the ETT | 2 hours
  defined as the mean of three readings of difference between inspiratory and expiratory tidal volumes (as measured by the anesthesia machine) at T0: after intubation, T1: immediately after recruitment, T2: 10 min after recruitment, T3: 20 min after recruitment, T4: at the end of surgery.
Number of attempts to insert and correctly size the tracheal tube. | 10 minutes
  Number of attempts to insert and correctly size the tracheal tube.
Desaturation incidence | 30 minutes postoperative
  (SPO2 less than 95%) at 1 min, 5 min, 10 min, 15 min, 20 min and 30 min postoperatively.
Hoarseness of voice. | 30 minutes postoperative
  Hoarseness of voice. Graded as follow:
  0= no hoarseness (good high-pitched cry sound)
  1. mild hoarseness (good cry but soft whispering low-pitched sound)
  2. severe hoarseness (cry but no audible sound)
Croup incidence | 30 minutes postoperative
  Croup (defined as triad of barking cough, stridor and a hoarse voice).

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarhan K, Walaa R, Hasanin A, Elgohary M, Alkonaiesy R, Nawwar K, Elsonbaty M, Elsonbaty A. Cuffed versus uncuffed endotracheal tubes in neonates undergoing noncardiac surgeries: A randomized controlled trial. Paediatr Anaesth. 2024 Oct;34(10):1045-1052. doi: 10.1111/pan.14953. Epub 2024 Jun 22. PMID 38922733